CLINICAL TRIAL: NCT05220995
Title: The Effects of Miminal Stimulation Protocol on Clinical Outcomes of Advanced Maternal Aged Women With Preimplantation Genetic Screening
Brief Title: The Effects of Miminal Stimulation Protocol on Preimplantation Genetic Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gokalp Oner (Other)
Responsible Party: Sponsor-Investigator, Gokalp Oner, Adem Yavuz, Nigde Omer Halisdemir University
Organization: Nigde Omer Halisdemir University (Other)
Other Study IDs: 31.01.2022
Record Dates: First submitted 2022-01-31; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Preimplantation Genetic Screening
Keywords: preimplantation genetic screening; gonadotropin dosage; euploidy rates
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — embryo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 100 patients with minimal: In advancing maternal age (AMA) women, minimal stimulation protocol (MSP) with the new combination of human menopausal gonadotrophin (hMG) and clomiphene citrate (CC) were performed for controlled ovarian hyperstimulation is defined for poor ovarian response women.
  Interventions: Genetic: protocol
- 100 patients with recombinant FSH antagonist protocol: In advancing maternal age (AMA) women, flexible antagonist protocol with recombinant FSH were performed for controlled ovarian hyperstimulation is defined for poor ovarian response women.
  Interventions: Genetic: protocol

INTERVENTIONS:
Genetic: protocol — ovarian stimulation protocols on euploid rates were compared.

SUMMARY:
PGS has been the most effective method for embryo selection in IVF cycles. Euploidy rates decrease significantly with advancing maternal age (AMA). The dosage of gonadotropins also may be increased to recruit an adequate number of follicles in AMA women, minimal Stimulation Protocol (MSP) with the new combination of human menopausal gonadotrophin (hMG) and clomiphene citrate (CC) for controlled ovarian hyperstimulation is defined for poor ovarian response women. The aim of this study is to show minimal stimulation protocol affect euploidy and pregnancy rates in preimplatation genetic screening (PGS) cycles with single embryo transfer.

ELIGIBILITY:
Inclusion Criteria: Advanced maternal aged -

Exclusion Criteria: Severe male factor, endometriosis, and absolute tubal factor were excluded in this study.

-

Ages: 38 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — more than 38 years old
Study Population: 200 advanced maternal aged women
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-01-23 (Estimated); Study Completion 2022-01-25 (Estimated)

PRIMARY OUTCOMES:
euploid rates | 3 months
  the effects of different stimulation protocols on euploid rates

SECONDARY OUTCOMES:
pregnancy rates | 3 months
  the effects of different stimulation protocols on pregnancy rates

CONTACTS AND LOCATIONS:
Locations (1):
- Gokalp Oner, Kayseri, Gevher Nesibe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We can not share.